CLINICAL TRIAL: NCT02379585
Title: A Pilot Study of Short-term Fasting on Neoadjuvant Chemotherapy in Patients With Newly Diagnosed Breast Cancer (STEFNE Study)
Brief Title: Fasting on Newly Diagnosed Breast Cancer
Acronym: STEFNE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI Decision
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1145332
Record Dates: First submitted 2015-01-12; First posted 2015-03-05 (Estimated); Results first posted 2017-11-08 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-03

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Doxorubicin; Cyclophosphamide; Enfuvirtide; Paclitaxel; Docetaxel; Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HER2 negative breast cancer (Active Comparator): Doxorubicin and cyclophosphamide every two weeks for four cycles (one cycle is defined as 14 days). After completing fourth cycle, paclitaxel every two weeks for an additional four cycles. The appropriate surgery will be done three to six weeks after completing the last cycle of paclitaxel.
  Interventions: Drug: Doxorubicin; Drug: cyclophosphamide; Drug: paclitaxel
- HER2 positive breast cancer (Active Comparator): Docetaxel, trastuzumab, and pertuzumab every three weeks for four cycles. Pegfilgrastim after docetaxel. Surgery three to six weeks after completing the last docatexel. If additional chemotherapy is needed patients will receive both doxorubicin and cyclophosphamide every three weeks for four cycles and after the fourth cycle then trastuzumab for one year
  Interventions: Drug: docetaxel; Drug: Trastuzumab; Drug: Pertuzumab

INTERVENTIONS:
Drug: Doxorubicin — doxorubicin (A) 60 mg/m2 plus cyclophosphamide (C) 600 mg/m2 every 2 weeks for four cycles followed by paclitaxel (T) 75 mg/m2 every 2 weeks for four cycles (dose-dense AC + T).20
  Other Names: (dose-dense AC + T).2
  Arms: HER2 negative breast cancer
Drug: cyclophosphamide — doxorubicin (A) 60 mg/m2 plus cyclophosphamide (C) 600 mg/m2 every 2 weeks for four cycles followed by paclitaxel (T) 75 mg/m2 every 2 weeks for four cycles (dose-dense AC + T).20
  Other Names: (dose-dense AC + T).20
  Arms: HER2 negative breast cancer
Drug: paclitaxel — For patients with HER2 negative breast cancer: doxorubicin (A) 60 mg/m2 plus cyclophosphamide (C) 600 mg/m2 every 2 weeks for four cycles followed by paclitaxel (T) 75 mg/m2 every 2 weeks for four cycles (dose-dense AC + T).20
  Other Names: (dose-dense AC + T).20
  Arms: HER2 negative breast cancer
Drug: docetaxel — For patients with HER2 positive breast cancer: docetaxel (T) 75 mg/m2 every 3 weeks for four cycles. Trastuzumab (H, 8mg/kg for 1st cycle, then 6 mg/kg in subsequent 3 cycles), Pertuzumab (P, 840 mg for 1st cycle, then 420 mg in subsequent 3 cycles) will be given concurrently with docetaxel for a total of 4 cycles before surgery. For patients who do not achieve pCR, adjuvant chemotherapy with doxorubicin (A) 60 mg/m2 plus cyclophosphamide (C) 600 mg/m2 every 3 weeks for four cycles will be given, followed by trastuzumab 6 mg/kg every 3 weeks to complete 1 year of treatment. For patients with pCR, only trastuzumab 6 mg/kg every 3 weeks will be given adjuvantly to complete 1 year of treatment (TPH + AC).21
  Other Names: (TPH + AC).21
  Arms: HER2 positive breast cancer
Drug: Trastuzumab — docetaxel (T) 75 mg/m2 every 3 weeks for four cycles. Trastuzumab (H, 8mg/kg for 1st cycle, then 6 mg/kg in subsequent 3 cycles), Pertuzumab (P, 840 mg for 1st cycle, then 420 mg in subsequent 3 cycles) will be given concurrently with docetaxel for a total of 4 cycles before surgery. For patients who do not achieve pCR, adjuvant chemotherapy with doxorubicin (A) 60 mg/m2 plus cyclophosphamide (C) 600 mg/m2 every 3 weeks for four cycles will be given, followed by trastuzumab 6 mg/kg every 3 weeks to complete 1 year of treatment. For patients with pCR, only trastuzumab 6 mg/kg every 3 weeks will be given adjuvantly to complete 1 year of treatment (TPH + AC).21
  Other Names: (TPH + AC).21
  Arms: HER2 positive breast cancer
Drug: Pertuzumab — docetaxel (T) 75 mg/m2 every 3 weeks for four cycles. Trastuzumab (H, 8mg/kg for 1st cycle, then 6 mg/kg in subsequent 3 cycles), Pertuzumab (P, 840 mg for 1st cycle, then 420 mg in subsequent 3 cycles) will be given concurrently with docetaxel for a total of 4 cycles before surgery. For patients who do not achieve pCR, adjuvant chemotherapy with doxorubicin (A) 60 mg/m2 plus cyclophosphamide (C) 600 mg/m2 every 3 weeks for four cycles will be given, followed by trastuzumab 6 mg/kg every 3 weeks to complete 1 year of treatment. For patients with pCR, only trastuzumab 6 mg/kg every 3 weeks will be given adjuvantly to complete 1 year of treatment (TPH + AC).21
  Other Names: (TPH + AC).21
  Arms: HER2 positive breast cancer

SUMMARY:
This study is to see how safe the use of short-term fasting is in breast cancer patients who will receive chemotherapy before undergoing surgery and to examine if the use of short-term fasting will decrease the side effects of chemotherapy and how much a tumor shrinks while receiving chemotherapy.

DETAILED DESCRIPTION:
Patients will fast 24 hours before and 24 hours after the administration of chemotherapy which will consist of doxorubicin plus cyclophosphamide every 2 weeks for four cycles followed by paclitaxel every 2 weeks for four cycles (dose-dense AC + T) or docetaxel (T) every 3 weeks for four cycles. Trastuzumab (H) and Pertuzumab (P) will be given concurrently with docetaxel for a total of 4 cycles before surgery. For patients who do not achieve pathological complete remission (pCR), adjuvant chemotherapy with doxorubicin (A) plus cyclophosphamide (C) every 3 weeks for four cycles will be given, followed by trastuzumab every 3 weeks to complete 1 year of treatment. For patients with pCR, only trastuzumab every 3 weeks will be given adjuvantly to complete 1 year of treatment (TPH + AC).

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age with histologically, and radiographically confirmed non-metastatic breast cancer with minimal tumor size over 1 cm (≥T1c lesion) to receive neoadjuvant chemotherapy recommended by the treating physician
* For estrogen receptor (ER) strongly positive, human epithelial receptor (HER2) negative breast cancer, Oncotype Dx study is required. Patients with low recurrence score will be excluded in the study.
* Eastern Cooperative Oncology Group (ECOG) performance status score < 1
* Absolute neutrophil count > 1500 mm3, platelet count ≥ 100×109 L, hemoglobin ≥ 8.5 g/dL
* Serum creatinine ≤1.5 times the upper limit of the normal range, total bilirubin ≤ 1.5 X ULN (≤ 3 mg/dL if clinically diagnosed with Gilbert syndrome) AST/ALT ≤ 2.5 X ULN (AST/ALT ≤ 5X ULN if clinically diagnosed with Gilbert syndrome)
* Willing to provide blood samples for correlative research purposes
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must be willing to use an acceptable contraceptive method (abstinence, oral contraceptive or double barrier method) for the duration of the study and for 30 days following the last dose of study drug, and must have a negative urine or serum pregnancy test within 2 weeks prior to beginning treatment on this trial.

Exclusion Criteria:

1. Uncontrolled cardiac disease, such as angina, hypertension or significant arrhythmias, congestive heart failure (NYHA grade 2 or more or LVEF < 40% on any prior assessment). Note: Assessment of LVEF is done before and after anthracycline-based or trastuzumab-based chemotherapy as standard of care
2. Pregnant or lactating females
3. Known history of diabetes mellitus. If screening fasting glucose is ≥126 mg/dL, an HbA1C must be < 6.5%.
4. History of syncope with calorie restriction in the past
5. Body mass index (BMI) < 19 kg/m2
6. Clinical signs or symptoms of GI obstruction and/or requirement for parenteral hydration or nutrition
7. Inability to complete informed consent process and adhere to the protocol treatment plan and follow-up requirements
8. Concurrent severe illness such as active infection, or psychiatric illness/social situations that would limit safety and compliance with study requirements
9. Any other medical comorbidity that requires daily medication(s) that may not be safely taken without food.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Waypa, FNP, Study Director — Research Director
Locations (1):
- Western Regional Medical Center, Goodyear, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnosed With HER2 Negative Breast Cancer: Patients will receive doxorubicin and cyclophosphamide every two weeks for four cycles (one cycle is defined as 14 days). After completing fourth cycle, they will receive paclitaxel every two weeks for an additional four cycles. The appropriate surgery will be done three-six weeks after completing the last cycle of paclitaxel.
  Doxorubicin: For patients with HER2 negative breast cancer: doxorubicin (A) 60 mg/m2 plus cyclophosphamide (C) 600 mg/m2 every 2 weeks for four cycles followed by paclitaxel (T) 75 mg/m2 every 2 weeks for four cycles (dose-dense AC + T).20
  cyclophosphamide: For patients with HER2 negative breast cancer: doxorubicin (A) 60 mg/m2 plus cyclophosphamide (C) 600 mg/m2 every 2 weeks for four cycles followed by paclitaxel (T) 75 mg/m2 every 2 weeks for four cycles (dose-dense AC + T).20
  paclitaxel: For patients with HER2 negative breast cancer: doxorubicin (A) 60 mg/m2 plus cyclophosphamide (C) 600 mg/m2 every 2 weeks for four cycles followed by paclitaxel (
- Diagnosed With HER2 Positive Breast Cancer: will receive docetaxel, trastuzumab, and pertuzumab every three weeks for four cycles (one cycle is defined as 21 days). An injection of pegfilgrastim will be administered after chemotherapy with docetaxel. The appropriate surgery will be done three to six weeks after completing the last cycle of docatexel. If the study doctor determines that additional chemotherapy is needed (based on tumor shrinkage), patients will receive both doxorubicin and cyclophosphamide every three weeks for four cycles and after the fourth cycle you will receive trastuzumab every three weeks for one year or patients will receive trastuzumab alone every three weeks for up to one year
  docetaxel: For patients with HER2 positive breast cancer: docetaxel 75 mg/m2 every 3 weeks for four cycles. Trastuzumab (H, 8mg/kg for 1st cycle, then 6 mg/kg in subsequent 3 cycles), Pertuzumab (P, 840 mg for 1st cycle, then 420 mg in subsequent 3 cycles) will be given concurrently with docetaxel for a total of 4 cycles be
Period: Overall Study
Arm/Group | Diagnosed With HER2 Negative Breast Cancer | Diagnosed With HER2 Positive Breast Cancer
Started | 3 | 5
Completed | 0 | 0
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Population: Data not collected. PI no longer at this institution
Groups:
- Diagnosed With HER2 Negative Breast Cancer: Patients will receive doxorubicin and cyclophosphamide every two weeks for four cycles (one cycle is defined as 14 days). After completing fourth cycle, they will receive paclitaxel every two weeks for an additional four cycles. The appropriate surgery will be done three to six weeks after completing the last cycle of paclitaxel.
- Diagnosed With HER2 Positive Breast Cancer: will receive docetaxel, trastuzumab, and pertuzumab every three weeks for four cycles (one cycle is defined as 21 days). An injection of pegfilgrastim will be administered after chemotherapy with docetaxel. The appropriate surgery will be done three to six weeks after completing the last cycle of docatexel. If the study doctor determines that additional chemotherapy is needed (based on tumor shrinkage), patients will receive both doxorubicin and cyclophosphamide every three weeks for four cycles and after the fourth cycle you will receive trastuzumab every three weeks for one year or patients will receive trastuzumab alone every three weeks for up to one year
- Total: Total of all reporting groups
Arm/Group | Diagnosed With HER2 Negative Breast Cancer | Diagnosed With HER2 Positive Breast Cancer | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Region of Enrollment

OUTCOME MEASURES:

1. Primary Outcome: Pathological Response Rate at the Time of Surgery or at the Time of Biopsy
Description: Evaluate pathological complete remission rate at the time of surgery, or partial pathological response rate (defined as residual invasive disease of 1cm) at the time of surgery or at the time of biopsy upon completion of planned chemotherapy.
Time Frame: 4-6 cycles (up to 12 weeks)
Population: Data not collected. The study has been terminated due to the PI no longer being employed at CTCA and not having rights to the trial information. After much effort, results were not able to be retained.
Arm/Group | Diagnosed With HER2 Negative Breast Cancer | Diagnosed With HER2 Positive Breast Cancer
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Fasting on the Toxicity of Neoadjuvant Chemotherapyaccording to the NCI
Description: The effect of short-term fasting on the toxicity of neoadjuvant chemotherapy in breast cancer patients according to the NCI common toxicity criteria (Version 4.03)
Time Frame: 4-6 cycles (up to 12 weeks)
Population: Data not collected. The study has been terminated due to the PI no longer being employed at CTCA and not having rights to the trial information."After much effort, results were not able to be retained.
Groups:
- Diagnosed With HER2 Negative Breast Cancer: Patients will receive doxorubicin and cyclophosphamide every two weeks for four cycles.
- Diagnosed With HER2 Positive Breast Cancer: Will receive docetaxel, trastuzumab, and pertuzumab every three weeks for four cycles (one cycle is defined as 21 days).
Arm/Group | Diagnosed With HER2 Negative Breast Cancer | Diagnosed With HER2 Positive Breast Cancer
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pathological Response Rate at the Time of Surgery or Time of Biopsy Upon Completion of Planned Chemotherapy
Description: To evaluate pathological complete remission rate (defined as disappearance of all invasive tumor in the breast; ypT0-is) at the time of surgery, or partial pathological response rate (defined as residual invasive disease of 1cm, ypT1a-b) at the time of surgery or at the time of biopsy upon completion of planned chemotherapy for triple-negative breast cancer.
Time Frame: 4-6 cycles
Population: as for outcome 2
Arm/Group | Diagnosed With HER2 Negative Breast Cancer | Diagnosed With HER2 Positive Breast Cancer
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Insulin Abnormalities
Description: Changes in plasma insulin abnormalities after short-term fasting and chemotherapy
Time Frame: 4-6 cycles (up to 12 weeks)
Population: as for outcome 2
Arm/Group | Diagnosed With HER2 Negative Breast Cancer | Diagnosed With HER2 Positive Breast Cancer
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Biomarker Changes Before and After Chemotherapy
Description: Biomarker changes in breast cancer (biopsy or residual tumor) before and after neoadjuvant chemotherapy
Time Frame: 4-6 cycles (up to 12 weeks)
Population: as for outcome 2
Arm/Group | Diagnosed With HER2 Negative Breast Cancer | Diagnosed With HER2 Positive Breast Cancer
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Nutritional Assessment Before and After Neoadjuvant Chemotherapy
Description: Nutritional status assessment with Patient Generated Subjective Global Assessment (aPG-SGA) before and after neoadjuvant chemotherapy
Time Frame: 4-6 cycles (up to 12 weeks)
Population: as for outcome 2
Arm/Group | Diagnosed With HER2 Negative Breast Cancer | Diagnosed With HER2 Positive Breast Cancer
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Glucose After Fasting and Chemotherapy
Description: To investigate changes in glucose after short-term fasting and chemotherapy
Time Frame: 4-6 cycles (up to 12 weeks)
Population: as for outcome 2
Arm/Group | Diagnosed With HER2 Negative Breast Cancer | Diagnosed With HER2 Positive Breast Cancer
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Changes in Insulin-like Growth Factor-1
Description: To investigate changes in Insulin-like growth factor-1 (IGF1) after short-term fasting and chemotherapy
Time Frame: 4-6 cycles (up to 12 weeks)
Population: as for outcome 2
Arm/Group | Diagnosed With HER2 Negative Breast Cancer | Diagnosed With HER2 Positive Breast Cancer
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Plasma Blood-based Tumor-related Abnormalities in DNA
Description: To investigate changes in plasma blood-based tumor-related abnormalities in DNA after short-term fasting and chemotherapy
Time Frame: 4-6 cycles (up to 12 weeks)
Population: as for outcome 2
Arm/Group | Diagnosed With HER2 Negative Breast Cancer | Diagnosed With HER2 Positive Breast Cancer
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: NA Data was not collected
Groups:
- Diagnosed With HER2 Negative Breast Cancer: Patients will receive doxorubicin and cyclophosphamide every two weeks for four cycles (one cycle is defined as 14 days). After completing fourth cycle, they will receive paclitaxel every two weeks for an additional four cycles. The appropriate surgery will be done three to six weeks after completing the last cycle of paclitaxel.
  0
Arm/Group | Diagnosed With HER2 Negative Breast Cancer | Diagnosed With HER2 Positive Breast Cancer
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes